CLINICAL TRIAL: NCT04632264
Title: Optimal Timing of Postpartum Oxytocin Administration in the Era of Delayed Cord Clamping - PROCEEDING (PostpaRtum OxytoCin Era dElayed corD clampING) Study
Brief Title: Postpartum Oxytocin Administration in the Era of Delayed Cord Clamping
Acronym: PROCEEDING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAS9154
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Two parallel randomized, placebo-controlled, and double-blinded studies. For this study we will include 52 scheduled cesarean sections and 52 vaginal deliveries as two separate cohorts.
Who Masked: Participant, Care Provider
Masking Description: Randomization will be achieved using a computer generated algorithm. Both patient and provider will be unaware of the allocation arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pre-placental group (Experimental): Oxytocin will be initiated immediately after delivery of the neonatal anterior shoulder (within 15 seconds). This is our "intervention" group. Saline placebo will be initiated post placenta delivery (within 15 seconds).
  Interventions: Other: Initiation of standard postpartum oxytocin immediately following fetal shoulder delivery; Other: Saline Placebo
- Post-placental group (Other): Saline placebo will be initiated post fetal shoulder delivery (within 15 seconds). Oxytocin will be initiated immediately after placenta delivery (within 15 seconds).
  Interventions: Other: Initiation of standard postpartum oxytocin immediately following placenta delivery; Other: Saline Placebo

INTERVENTIONS:
Other: Initiation of standard postpartum oxytocin immediately following fetal shoulder delivery — The intervention is to determine if initiating oxytocin as soon as the fetus is delivered decreased postpartum blood loss. 30 units in 500 milliliters of 0.9% sodium chloride
  Arms: Pre-placental group
Other: Initiation of standard postpartum oxytocin immediately following placenta delivery — Standard of care includes oxytocin administration post-delivery regardless of delivery mode. This is the comparative group. 30 units in 500 milliliters of 0.9% sodium chloride
  Arms: Post-placental group
Other: Saline Placebo — Saline placebo will be initiated post placenta delivery (within 15 seconds).
  Arms: Pre-placental group
Other: Saline Placebo — Saline placebo will be initiated post fetal shoulder delivery (within 15 seconds).
  Arms: Post-placental group

SUMMARY:
Increased blood loss after vaginal or cesarean delivery is one of the top causes of maternal complications. Oxytocin is a common medication given to mothers by IV or an injection to limit the amount of blood loss after delivery. The investigators do not know the best time after delivery that oxytocin should be given. This research is being done to find out if starting the medication oxytocin right after the baby is born or after the placenta comes out decreases the amount of blood lost after birth when we delay cord clamping after birth.

DETAILED DESCRIPTION:
The optimal timing of prophylactic oxytocin administration on both maternal and neonatal outcomes has not been definitively established with delayed cord clamping. Maternal considerations include the risk of postpartum hemorrhage, need for additional uterotonic medications, need for maternal transfusion, retained placenta, and postpartum drop in hemoglobin. Neonatal considerations include markers of neonatal well-being such as arterial pH and 5-minute Apgar score, as well as hemoglobin and bilirubin levels. There is currently no protocol on the timing of third stage prophylactic oxytocin and its administration is based on physician/ delivery provider's preference. The investigators propose a quality assessment initiative, through a randomized controlled trial designed to compare the blood loss between administrations of prophylactic oxytocin immediately after delivery of the neonate versus after delivery of the placenta with delayed cord clamping.

ELIGIBILITY:
Inclusion Criteria:

* All laboring women (induced, augmented, or spontaneous) at term admitted to Labor and Delivery while comfortable
* Scheduled cesareans
* Women aged 18 years or older
* Admitted at NewYork-Presbyterian Morgan Stanley Children's Hospital (CHONY) or Allen Pavilion Labor and Delivery units

Exclusion Criteria:

* Multifetal gestation
* Placental abruption or antepartum hemorrhage
* Maternal bleeding disorder
* Known fetal anomaly or anemia
* Fetal growth restriction with abnormal Doppler
* Significant maternal anemia (pre-operative hemoglobin ≤ 7g/dL
* Intrapartum stillbirth
* Placenta accreta spectrum
* Abnormal placentation (previa or abruption)
* Planned cord blood banking
* Refusal of blood products
* Any contraindication for delayed cord clamping
* Maternal history of aortic stenosis or pulmonary hypertension or other severe cardiac structural disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin | Up to 24 hours
  Change defined as greater or equal to 1.0 g/dL (≥ 1 standard deviation (SD)) hemoglobin drop between the two arms following a vaginal delivery and greater or equal to 0.9 g/dL (≥ 1SD) following a cesarean delivery.

SECONDARY OUTCOMES:
Cumulative Maternal Adverse Outcomes | Postpartum, Up to 6 weeks
  Any adverse maternal outcome (adverse event) including blood transfusion or symptomatic anemia.
Cumulative Neonatal Adverse Outcomes | Post Delivery, Up to 6 weeks
  Any adverse neonatal outcome (adverse event) including jaundice, hematocrit laboratory abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E. Purish, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Soltani H, Hutchon DR, Poulose TA. Timing of prophylactic uterotonics for the third stage of labour after vaginal birth. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD006173. doi: 10.1002/14651858.CD006173.pub2. PMID 20687079
- [Background] GBD 2015 Maternal Mortality Collaborators. Global, regional, and national levels of maternal mortality, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1775-1812. doi: 10.1016/S0140-6736(16)31470-2. PMID 27733286
- [Background] Rana N, Kc A, Malqvist M, Subedi K, Andersson O. Effect of Delayed Cord Clamping of Term Babies on Neurodevelopment at 12 Months: A Randomized Controlled Trial. Neonatology. 2019;115(1):36-42. doi: 10.1159/000491994. Epub 2018 Oct 2. PMID 30278462
- [Background] Andersson O, Lindquist B, Lindgren M, Stjernqvist K, Domellof M, Hellstrom-Westas L. Effect of Delayed Cord Clamping on Neurodevelopment at 4 Years of Age: A Randomized Clinical Trial. JAMA Pediatr. 2015 Jul;169(7):631-8. doi: 10.1001/jamapediatrics.2015.0358. PMID 26010418
- [Background] Andersson O, Hellstrom-Westas L, Andersson D, Domellof M. Effect of delayed versus early umbilical cord clamping on neonatal outcomes and iron status at 4 months: a randomised controlled trial. BMJ. 2011 Nov 15;343:d7157. doi: 10.1136/bmj.d7157. PMID 22089242
- [Background] Committee Opinion No. 684: Delayed Umbilical Cord Clamping After Birth. Obstet Gynecol. 2017 Jan;129(1):1. doi: 10.1097/AOG.0000000000001860. PMID 28002310
- [Background] Purisch SE, Ananth CV, Arditi B, Mauney L, Ajemian B, Heiderich A, Leone T, Gyamfi-Bannerman C. Effect of Delayed vs Immediate Umbilical Cord Clamping on Maternal Blood Loss in Term Cesarean Delivery: A Randomized Clinical Trial. JAMA. 2019 Nov 19;322(19):1869-1876. doi: 10.1001/jama.2019.15995. PMID 31742629
- [Background] Hamm RF, Wang EY, Bastek JA, Srinivas SK. Assessing reVITALize: Should the Definition of Postpartum Hemorrhage Differ by Mode of Delivery? Am J Perinatol. 2017 Apr;34(5):503-507. doi: 10.1055/s-0036-1593535. Epub 2016 Oct 12. PMID 27732984
- [Background] Jackson KW Jr, Allbert JR, Schemmer GK, Elliot M, Humphrey A, Taylor J. A randomized controlled trial comparing oxytocin administration before and after placental delivery in the prevention of postpartum hemorrhage. Am J Obstet Gynecol. 2001 Oct;185(4):873-7. doi: 10.1067/mob.2001.117363. PMID 11641669